CLINICAL TRIAL: NCT04755920
Title: A Feasibility Study of SGM-101, a Fluorochrome-labeled Anti-carcinoembryonic Antigen Monoclonal Antibody for the Intraoperative Detection of Colorectal Brain Metastases.
Brief Title: SGM-101 in Colorectal Brain Metastases.
Acronym: SGM-CBM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Medical Center Haaglanden (Other); Surgimab (Industry)
Responsible Party: Principal Investigator, Alexander Vahrmeijer, Oncologic Surgeon - Hepatobiliary and Colorectal, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL74956.058.20
Record Dates: First submitted 2021-01-27; First posted 2021-02-16 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Rectal Neoplasms; Rectum Cancer; Colorectal Neoplasms; Brain Metastases; Brain Neoplasms; Brain Diseases; Brain Cancer; Brain Tumor; Intestinal Neoplasms; Gastrointestinal Neoplasms; Gastrointestinal Cancer; Gastrointestinal Disease; Intestinal Disease
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms; Brain Neoplasms; Brain Diseases; Intestinal Neoplasms; Gastrointestinal Neoplasms; Gastrointestinal Diseases; Intestinal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with colorectal brain metastases (Experimental): 10 mg SGM-101, administration 3 to 5 days prior to surgery.
  Interventions: Drug: SGM-101

INTERVENTIONS:
Drug: SGM-101 — Fluorescence-guided surgery

SUMMARY:
This study assesses the feasibility of SGM-101, a fluorochrome-labeled anti-carcinoembryonic antigen monoclonal antibody, for intraoperative near-infrared fluorescence imaging of colorectal brain metastases by injecting SGM-101 intravenously 3 - 5 days prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure;
2. Patients aged over 18 years old;
3. All women of child bearing potential and all males must practice effective contraception during the study and be willing and able to continue contraception for at least 30 days after their last dose of study treatment.
4. Has the ability to communicate well with the Investigator in the Dutch language and willing to comply with the study restrictions.
5. Diagnosed with brain metastasis of colorectal origin and scheduled for a resection.

Exclusion Criteria:

1. History of any anaphylactic reaction;
2. Previous use of SGM-101;
3. Other malignancies either currently active or diagnosed in the last 5 years, except adequately treated in situ carcinoma of the cervix and basal or squamous cell skin carcinoma;
4. Laboratory abnormalities defined as:

   1. Aspartate AminoTransferase, Alanine AminoTransferase, Gamma Glutamyl Transferase) or Alkaline Phosphatase levels above 5 times the or;
   2. Total bilirubin above 2 times the ULN or;
   3. Serum creatinine above 1.5 times the ULN or;
   4. Platelet count below 100 x 109/L or;
   5. Hemoglobin below 4 mmol/L (females) or below 5 mmol/l (males);
   6. Known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) or hepatitis C virus (HCV) antibody or patients with untreated serious infections;
5. Patients pregnant or breastfeeding;
6. Any condition that the investigator considers to be potentially jeopardizing the patient's well-being or the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of SGM-101 for intraoperative imaging of colorectal brain metastases. | Intraoperative
  * Concordance between the fluorescent signal and the tumor status (incl. degree of CEA-expression) of resected tissue;
  * Concordance between the fluorescent signal and the resection margin with the use of neuronavigation

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Medical Center Haaglanden, The Hague

IPD SHARING:
Plan to Share IPD: No